CLINICAL TRIAL: NCT06343831
Title: Quantitative Assessment of Autologous Fat Transfer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Houston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB23-1646
Record Dates: First submitted 2024-03-05; First posted 2024-04-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Autologous Fat Grafting

STUDY DESIGN:
Intervention Model Description: Patients planning to undergo autologous fat transfer for breast or chest wall reconstruction will be enrolled prospectively. Participants will undergo standard photographs (2-D imaging) of their chest wall and torso, including the breasts, and complete a validated questionnaire (BREAST-QTM) to evaluate patient satisfaction, and quality of life, all standard of care. The 3D photographs, MRI, and US are routinely used in practice but will be performed for research purposes in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients Receiving Autologous Fat Transfer of the Breast or Chest Wall (Experimental): Participants will undergo standard photographs (2-D imaging) of their chest wall and torso, including the breasts, and complete a validated questionnaire (BREAST-QTM) to evaluate patient satisfaction, and quality of life, all standard of care. The 3D photographs, MRI, and US are routinely used in practice but will be performed for research purposes in this study.
  Interventions: Procedure: 2-Dimensional (2-D) Photographs (Visit 1/ Follow up Visit 3-6); Procedure: 3-Dimensional (3-D) Photographs (Visit 1- 6); Procedure: Ultrasound Soft Tissue Assessment (Visit 1/ Follow up Visit 4-6); Procedure: Magnetic Resonance Imaging Volume Assessment (Visit 1/ Follow up Visit 4-6); Procedure: BREAST-QTM questionnaire (Visit 1/ Follow up Visit 4-6)

INTERVENTIONS:
Procedure: 2-Dimensional (2-D) Photographs (Visit 1/ Follow up Visit 3-6) — The study participant will be requested to stand upright with hands comfortably behind their back and turn 45 degrees and 90 degrees in either direction for standard anteroposterior (AP), oblique and lateral photos. Standardized photographic poses will be utilized so that only the participant's neck and torso will be visible and all jewelry on the neck and arms will be removed to eliminate potential identifiers. The photographs will be acquired using a commercially available camera or study iPad device.
Procedure: 3-Dimensional (3-D) Photographs (Visit 1- 6) — 3-Dimensional surface scans of the participant's torso will be acquired using a commercially available handheld camera scanning device that offers texture, geometry, and color acquisition from any complex surface using white light technology, which is safe for exposure to skin and eyes. Prior to imaging, a pattern of lines and dots will be marked on the patient's breasts using a washable marker. The study participant will be requested to sit upright on the exam room table with hands comfortably behind their back while the research staff member moves around their torso with the handheld scanner. The exam room table will then be reclined to a lay-flat position such that the patient is laying supine, and breast imaging will be repeated. Standardized photographic poses will be utilized so that only the participant's neck and torso will be visible and all jewelry on the neck and arms will be removed to eliminate potential identifiers.
Procedure: Ultrasound Soft Tissue Assessment (Visit 1/ Follow up Visit 4-6) — The images will be acquired using a commercially available handheld ultrasound scanning device. The study participant will be requested to sit upright on the exam room table with hands comfortably behind their back while the research staff member obtains images of the specific area of the breast of chest wall to be grafted (V1) and that which was grafted (V4-6). Images usually take 5-10 minutes to acquire depending on the number of areas grafted.
Procedure: Magnetic Resonance Imaging Volume Assessment (Visit 1/ Follow up Visit 4-6) — An MRI of the breast will be obtained around visit 1 and visits 4-6 timepoints. The images will be acquired in collaboration with the Breast Imaging Core and the Magnetic Resonance Research Imaging Center. Dr. Abe (co-investigator, radiology) will review the images to assess volume of the overall breast, the specific areas of the breasts that were grafted.
Procedure: BREAST-QTM questionnaire (Visit 1/ Follow up Visit 4-6) — The BREAST-QTM measures three satisfaction domains and three quality of life (QoL) domains.6 For BREAST-QTM, each domain has a score range from 0 - 100. A difference in score, either positive or negative, of 10 points is considered clinically "important"; a difference of 20 points is considered clinically "very important." This survey will be administered to participants via iPad during visit 1 and visits 4-6 and takes approximately 10-20 minutes to complete.

SUMMARY:
This is a single-arm, prospective pilot study that will objectively assess outcomes in patients electively undergoing Autologous Fat Transfer (AFT) for breast or chest wall reconstruction. Patients planning to undergo autologous fat transfer for breast or chest wall reconstruction will be enrolled prospectively. Participants will undergo standard photographs (2-D imaging) of their chest wall and torso, including the breasts, and complete a validated questionnaire (BREAST-QTM) to evaluate patient satisfaction, and quality of life, all standard of care. The 3D photographs, Magnetic resonance imaging (MRI), and Ultrasound (US) are routinely used in practice but will be performed for research purposes in this study. All imaging procedures and questionnaires will be obtained at baseline and follow-up visits 3-6.

DETAILED DESCRIPTION:
The purpose of this pilot study is to assess the utility of imaging (photographs, ultrasound (US), and Magnetic resonance imaging (MRI) )to follow outcomes of autologous fat grafting to the chest for reconstruction. The study team will compare images obtained from each of these methods (photographs, ultrasound, and MRI) to visualize changes in the breast over time.

All participants will meet with a member of the research staff at a pre-operative appointment in the Center for Reconstructive Surgery. At Visit 1 participants will be consented, undergo research-specific data collection, surveys, US, MRI scan, 2D photographs, and 3D surface scanning of their torso/breast.

During follow-up Visits 3-6, participants will undergo research-specific 2D photographs and 3D surface scanning of their breast and chest wall. Participants will also have an ultrasound and MRI scan performed during follow-up visits 4-6 in addition to completing a questionnaire to evaluate patient satisfaction and quality of life following fat grafting.

After obtaining a Data Use Agreement (DUA), de-identified photographs and 3D scans of the participants' torsos (area of fat grafting) will be shared with the University of Houston (Dr. Fatima Merchant) to analyze using software developed to look specifically at volume of the breast before and after surgery and compare the 3D photos with the MRI data. No protected health information (PHI) will be shared with the University of Houston or other investigators.

During each clinic visit, relevant data will be extracted from Epic and entered manually into REDCap data forms by a member of the research team.

ELIGIBILITY:
Inclusion Criteria:

Age of 18 years or older

* Planned autologous fat transfer or fat grafting reconstruction of the breast or chest wall.
* Able to provide written or electronic informed consent.
* Able to undergo MRI.

Exclusion Criteria:

* Vulnerable subjects (children, prisoners, pregnant women).
* Patients who have active cancer, metastatic disease, solid organ transplantation / immunosuppression, or autoimmune diseases.
* Unable to undergo MRI (history of metal contraindication, claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in breast/chest wall following autologous fat grafting, measured by imaging. | Visit 1through study completion, an average of 1 year
  Images will be obtained from photographs, ultrasound, and MRI to compare and follow outcomes of autologous fat grafting to the chest for reconstruction and to visualize changes in the breast over time.

SECONDARY OUTCOMES:
Change from baseline in quality of life as measured by the BREAST-QTM survey. | Visit 1through study completion, an average of 1 year.
  The BREAST-QTM is utilized to assess patient- reported cosmetic and reconstructive breast surgery and clinical practice satisfaction and quality of life outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Summer Hanson, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - The University of Chicago, Chicago, Illinois
  - The University of Houston, Houston, Texas